CLINICAL TRIAL: NCT00332189
Title: A Phase 3b, Multicenter, Open-Label Extension Study of Phenoptin in Subjects With Phenylketonuria Who Participated in Protocols PKU-004 or PKU-006
Brief Title: Study of Phenoptin in Subjects With Phenylketonuria Who Participated in Protocols PKU-004 or PKU-006
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-008
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-10

CONDITIONS: Phenylketonuria
Keywords: PKU
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

INTERVENTIONS:
Drug: sapropterin dihydrochloride — 5-20mg/kg/day orally, dose may be adjusted up or down as needed at the discretion of the investigator in increments of 5mg/kg/day.
  Other Names: Kuvan

SUMMARY:
The objective of this study is to evaluate the safety of long-term treatment with Phenoptin in subjects with phenylketonuria (PKU) who participated in Phase 3 clinical studies with Phenoptin.

ELIGIBILITY:
Inclusion Criteria:

* Participation in study PKU-004 or PKU-006
* Willing and able to provide written, signed informed consent or, in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures
* Negative urine pregnancy test at screening (females of child-bearing potential)
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Non-responsive to prior treatment with Phenoptin based on participation in PKU-004 or PKU-006
* Perceived to be unreliable or unavailable for study participation or, if under the age of 18 years, have parents or legal guardians who are perceived to be unreliable or unavailable
* Terminated early from PKU-004 or PKU-006, except for subjects in PKU-004 that rolled into PKU-008 at Week 22, subjects in PKU-006 that rolled into PKU-008 at Week 10, or subjects in PKU-006 that terminated due to elevated Phe levels following dietary Phe increases
* Use of any investigational product other than Phenoptin within 30 days prior to screening, or anticipated requirement for any investigational agent prior to completion of all scheduled study assessments
* Positive urine pregnancy test at screening (non-sterile females of child-bearing potential only), already known to be pregnant or breastfeeding or planning a pregnancy in self or partner during the study
* Female subjects of childbearing potential must be using an effective method of birth control, as determined by the PI, and willing to continue to use acceptable birth control measures
* Concurrent disease or condition that would interfere with study participation or safety (e.g., seizure disorder, oral steroid-dependent asthma or other condition requiring oral or parenteral corticosteroid administration, or insulin-dependent diabetes)
* Any condition that, in the view of the PI, renders the subject at high risk from treatment compliance and/or completing the study
* ALT > 2 times the upper limit of normal (i.e., Grade 1 or higher based on World Health Organization Toxicity Criteria) at screening (see Appendix 2)
* Serious neuropsychiatric illness (e.g., major depression) not currently under medical control
* Prior history of organ transplantation
* Requirement for concomitant treatment with any drug known to inhibit folate synthesis (e.g., methotrexate)
* Concurrent use of levodopa
* Clinical diagnosis of primary BH4 deficiency

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Los Angeles, California
  - Sacramento, California
  - San Jose, California
  - New Haven, Connecticut
  - Atlanta, Georgia
  - Chicago, Illinois
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Portland, Oregon
  - Dallas, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Madison, Wisconsin

REFERENCES:
- [Derived] Burton BK, Nowacka M, Hennermann JB, Lipson M, Grange DK, Chakrapani A, Trefz F, Dorenbaum A, Imperiale M, Kim SS, Fernhoff PM. Safety of extended treatment with sapropterin dihydrochloride in patients with phenylketonuria: results of a phase 3b study. Mol Genet Metab. 2011 Aug;103(4):315-22. doi: 10.1016/j.ymgme.2011.03.020. Epub 2011 Mar 31. PMID 21646032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects had to have previously participated in study PKU-004 (NCT00225615) or PKU-006 (NCT00272792)
Pre-assignment Details: The last assessment obtained in PKU-004 or PKU-006 could be used to determine eligibility for this study provided assessment was conducted fewer than six weeks prior to PKU-008 Day 1.
Groups:
- Total Patient Population: Phenoptin will be taken orally once daily as the number of tablets equivalent to that of the last prescribed dose of the previous study (PKU-004 NCT00225615 or PKU-006 NCT00272792). Subjects who participated in PKU-006 NCT00272792 will receive Phenoptin as the number of tablets equivalent to 20 mg/kg/day at enrollment. The Phenoptin dose may be adjusted up or down as needed at the discretion of the investigator in increments of approximately 5 mg/kg/day within a range of 5 mg/kg/day to 20 mg/kg/day to control blood Phe to levels consistent with local clinical site recommendations for blood Phe control.
Period: Overall Study
Arm/Group | Total Patient Population
Started | 111
Completed | 90 (Subjects in this extension study continued until there was market approval in their region.)
Not Completed | 21
Not completed — Adverse Event | 3
Not completed — Uncooperative/Noncompliant | 3
Not completed — Withdrawal by Subject | 9
Not completed — Lack of Efficacy | 4
Not completed — Moved out of country | 2

BASELINE CHARACTERISTICS:
Groups:
- Total Patient Population: The mean (+/- SD) daily dose of study drug was 16.4 (+/-4.4) mg/kg. The final dose prescribed was 20 mg/kg/day for 73 (65.8%) subjects, 10 mg/kg/day for 33 (29.7%) subjects, and 5 mg/kg/day for 5 (4.5%) subjects.
Arm/Group | Total Patient Population
Number analyzed (Participants) | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 16.4 (10.2)
Age, Customized [Number; unit: participants]
  >=4 to <8 | 20
  >=8 to <12 | 24
  >=12 to <18 | 28
  >=18 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 67
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 108
  Asian/Asian Pacific Islander | 1
  Hispanic | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  North America | 54
  Europe | 57

OUTCOME MEASURES:

1. Primary Outcome: Tabulation of the Incidence and Frequency of All AEs and SAEs That Occur Throughout the Study.
Description: Safety was assessed with regards to the rate and type of AEs, clinically significant changes to vital signs and/or physical examination findings, and clinically significant changes in laboratory test results.
Time Frame: Baseline through Final Visit (a Maximum of 30 months) with AEs collected at month 3 and 6 then at 6 month intervals
Population: Percentage of total population who experienced an AE or SAE presented here. For full list of SAEs, and AEs experienced with a frequency of greater than 5%, see the Reported Adverse Event section.
Measure: Number; unit: percentage of subjects reporting events
Groups:
- Total Patient Population: The safety analysis population includes all subjects who received at least one dose of study drug during the study.
Arm/Group | Total Patient Population
Number analyzed (Participants) | 111
percentage of subjects reporting events
  % of Subjects Reporting Any Adverse Event | 83.8
  % of Subjects Reporting Related Adverse Events | 33.3
  % of Subjects Reporting Serious Adverse Events | 6.3
  % of Subjects Reporting Related Serious AEs | 0.9

2. Secondary Outcome: Following Blood Phe Levels.
Description: There were no pre-specified efficacy analysis, blood Phe samples were taken at each visit. Blood Phe concentrations remained within levels consistent with local clinical site recommendations for blood Phe control.
Time Frame: Baseline through Final Visit (a Maximum of 30 months) with blood phe samples taken at months 3 and 6 then at 6 month intervals
Population: The population includes all subjects who received at least one dose of study drug during the study and had at least one measurement of blood Phe level.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Total Patient Population
Number analyzed (Participants) | 111
micromoles per liter
  Baseline Blood Phe Level (N=111) | 607.4 (328.44)
  Month 3 Blood Phe Level (N=109) | 504.6 (316.33)
  Month 3 Change from Baseline (N=109) | -105.7 (287.20)
  Month 6 Blood Phe Level (N=104) | 529.9 (332.45)
  Month 6 Change from Baseline (N=104) | -68.0 (310.76)
  Month 12 Blood Phe Level (N=97) | 494.4 (330.57)
  Month 12 Change from Baseline (N=97) | -95.7 (304.81)
  Month 18 Blood Phe Level (N=58) | 526.9 (357.43)
  Month 18 Change from Baseline (N=58) | -92.8 (306.02)
  Month 24 Blood Phe Level (N=45) | 482.0 (322.55)
  Month 24 Change from Baseline (N=45) | -122.2 (281.03)
  Month 30 Blood Phe Level (N=1) | 808.0 (NA) — There was only one subject that had a 30 month visit.
  Month 30 Change from Baseline (N=1) | 542.0 (NA) — There was only one subject that had a 30 month visit.

ADVERSE EVENTS:
Time Frame: Maximum exposure to study drug was 953 days (2.6 years), with a median duration of 595.0, and a mean (+/- SD) duration of exposure of 658.7 (+/-221.3) days.
Arm/Group | Total Patient Population
Serious Adverse Events (participants affected / at risk) | 7/111
Other Adverse Events (participants affected / at risk) | 93/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Patient Population (N=111)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) — A 15 year old female who had perviously participated in PKU-001, PKU-003, and PKU-004, was taking Ibuprofen in addition to 7.2 mg/kg/day of sapropterin dihydrochloride. It is possible that this combination lead to the event of gastroesophageal reflux
Testicular mass (Reproductive system and breast disorders) | 1 (1) — The Investigator assessed this event as not related to study drug. The AE verbatim terms for this subject included, testicular mass, and lymphadenectomy.
Tonsillectomy (Surgical and medical procedures) | 1 (1) — The Investigator assessed the event as not related to study drug. The AE verbatim term for this subject was tonsilectomy.
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) — The Investigator assessed the event as not related to study drug. The AE verbatim term for this subject was menorrhagia and dysmenorrhoea.
Road traffic accident (Injury, poisoning and procedural complications) | 1 (2) — The Investigator assessed the event as not related to study drug. The AE verbatum terms for this subject included, upper back pain following road traffic accident, and neck pain following road traffic accident.
Hand Fracture (Injury, poisoning and procedural complications) | 1 (2) — The Investigator assessed this event as not related to study drug. The AE verbatim terms for this subject included, dislocation of left scapulo - humeral, fracture right hand, and fracture 3rd hand metacarpal and 4th basal metacarpal right hand.
Surgery (Surgical and medical procedures) | 1 (1) — The Investigator assessed the event as not related to study drug. The AE verbatim term for this subject was incontinence.
Lymphadenectomy (Surgical and medical procedures) | 1 (1) — The Investigator assessed this event as not related to study drug. The AE verbatim terms for this subject included, testicular mass, and lymphadenectomy.
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) — The Investigator assessed this event as not related to study drug. The AE verbatim terms for this subject included, dislocation of left scapulo - humeral, fracture right hand, and fracture 3rd hand metacarpal and 4th basal metacarpal right hand.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Patient Population (N=111)
Bronchitis (Infections and infestations) | 6 (7) — Events listed in the Other Adverse Events Table include events assessed as related to study drug and events assessed as non-related to study drug.
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (28)
Diarrhoea (Gastrointestinal disorders) | 10 (16)
Gastroenteritis (Infections and infestations) | 7 (7)
Gastroenteritis viral (Infections and infestations) | 8 (9)
Headache (Nervous system disorders) | 13 (48)
Influenza (Infections and infestations) | 9 (15)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Nasopharyngitis (Infections and infestations) | 20 (30)
Pharyngitis (Infections and infestations) | 7 (13)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (15)
Pyrexia (General disorders) | 18 (25)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 22 (28)
Viral infection (Infections and infestations) | 8 (12)
Vomiting (Gastrointestinal disorders) | 20 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the results shall be made in a joint publication. If such a multi-center publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from their site individually, subject however, to compliance with the other terms of the agreement.